CLINICAL TRIAL: NCT02223234
Title: Guelph Family Health Study: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Jess Haines, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14AP008
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Control- monthly mailed information on children's health
  Interventions: Behavioral: Control
- Email and 4 Home Visits (Experimental): Weekly emails and 4 home visits with a health educator
  Interventions: Behavioral: Emails and 4 Home Visits
- Email and 2 Home Visits (Experimental): Weekly emails and 2 home visits
  Interventions: Behavioral: Emails and 2 home visits

INTERVENTIONS:
Behavioral: Emails and 4 Home Visits — Weekly emails and 4 home visits with health educator
  Arms: Email and 4 Home Visits
Behavioral: Control — Monthly emails on child health
  Arms: Control
Behavioral: Emails and 2 home visits — Weekly emails and 2 home visits with health educator
  Arms: Email and 2 Home Visits

SUMMARY:
The overall objective of the proposed study is to test, among Canadian families, the comparative effectiveness of 2 different versions (doses) of a family-based obesity prevention intervention that is tailored to families' behavioural risk profile.

To achieve this objective, we will conduct a randomized controlled trial of families with children aged 18 months- 5 years. Families will be randomized to 1 of 3 conditions: 1) Monthly emails with general health information (Attention Control), 2) Tailored weekly emails and 2 home visits with a health educator (Email +2), 3) Tailored weekly emails and 4 home visits (Email +4). The intervention will last 6 months, with follow-up at 12-months post-intervention (18 months from baseline). We will examine the impact of the intervention on the children's body composition, weight-related behaviours, and biomarkers of diabetes and cardiovascular disease risk.

We hypothesize that, compared to children in the Attention Control, children in the Email +2 and Email +4 conditions will achieve:

1. a smaller increase in adiposity (primary outcome), age- and gender-specific body mass index (BMI),over a 6-month intervention period.
2. higher frequency of family meals, child's sleep duration, physical activity, and fruit and vegetable intake and lower child's sugar-sweetened beverage intake, and sedentary behaviour over a 6-month intervention period. (secondary outcomes)
3. lower diastolic blood pressure, glycosylated hemoglobin, fasting glucose, fasting insulin, Low Density Lipoprotein (LDL) cholesterol, triglycerides, C-reactive protein, trans and saturated fats, and higher High Density Lipoprotein (HDL) cholesterol over a 6-month intervention period.

We further hypothesize that there will be no significant difference in these outcomes between children in the conditions with 2 (Email +2) or 4 (Email +4) home visits.

ELIGIBILITY:
Inclusion Criteria:

* families who have a child aged 18 months through 5 years
* live the Guelph area
* have a parent who can respond to questionnaires in English

Exclusion Criteria:

* families who plan to move during the study period
* children with severe health conditions (such as severe cerebral palsy) that would prohibit them from participating in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change in adiposity | baseline, 6 month follow-up

SECONDARY OUTCOMES:
change in body mass index | baseline, 6-month follow-up
change in waist circumference | baseline, 6-month follow-up
change in frequency of family meals | baseline, 6-month follow-up
change in child's sleep duration | baseline, 6-months
change in child's physical activity | baseline, 6-months
change in child's fruit and vegetable intake | baseline, 6-month follow-up
change in child's sugar-sweetened beverage intake | baseline, 6-month follow-up
change in sedentary behaviour | baseline, 6-month follow-up
change in child's diastolic blood pressure | baseline, 6-month follow-up
change in child's biomarkers of diabetes and cardiovascular disease risk | baseline, 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Krystia O, Ambrose T, Darlington G, Ma DWL, Buchholz AC, Haines J; Guelph Family Health Study. A randomized home-based childhood obesity prevention pilot intervention has favourable effects on parental body composition: preliminary evidence from the Guelph Family Health Study. BMC Obes. 2019 Mar 4;6:10. doi: 10.1186/s40608-019-0231-y. eCollection 2019. PMID 30873285
- [Derived] Haines J, Douglas S, Mirotta JA, O'Kane C, Breau R, Walton K, Krystia O, Chamoun E, Annis A, Darlington GA, Buchholz AC, Duncan AM, Vallis LA, Spriet LL, Mutch DM, Brauer P, Allen-Vercoe E, Taveras EM, Ma DWL; Guelph Family Health Study. Guelph Family Health Study: pilot study of a home-based obesity prevention intervention. Can J Public Health. 2018 Aug;109(4):549-560. doi: 10.17269/s41997-018-0072-3. Epub 2018 Apr 25. PMID 29981086